CLINICAL TRIAL: NCT05218174
Title: Exercise Training and Functional, Cognitive, and Emotional Well-being in Adults with Post-Acute Sequelae of SARS-CoV-2 (COVID-19) Infection (PASC): a Randomized Controlled Trial
Brief Title: Exercise in Adults with Post-Acute Sequelae of SARS-CoV-2 (COVID-19) Infection Study
Acronym: PASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Sports Academy (Unknown)
Responsible Party: Principal Investigator, Simon Driver, Research Center Director - The STAR at Frisco, Baylor Research Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 021-347
Record Dates: First submitted 2021-11-22; First posted 2022-02-01 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise training program (Experimental): Participants in this arm will complete an 8-week exercise training program comprised of an initial functional assessment to create an exercise prescription, followed by 7 in-person weekly sessions. Each session consisting of approximately 50 minutes of individualized exercise training and approximately 10 minutes of cognitive training via the Sports Academy "CogPT" iPad app. All participants will receive exercise and cognitive training delivered weekly in a group-based setting at Sports Academy within the Star in Frisco, Texas during the intervention period. Additionally, they will have access to daily workouts pushed to their phone via the MOVE exercise app developed by our team.
  Interventions: Other: Exercise Prescription
- No training program (Sham Comparator): Participants in this arm will be wearing the WHOOP band for 8-weeks but will not be exposed to any active intervention.
  Interventions: Other: Exercise Prescription

INTERVENTIONS:
Other: Exercise Prescription — In this prospective, randomized control trial, the investigators will compare functional exercise capacity, cognitive performance, and emotional well-being at baseline and following 2 conditions: (1) an 8-week exercise training program (intervention) or (2) no training program (control). Participants will be randomized using a 1:1 randomization scheme into either the intervention or control group. After 8 weeks, participants in the wait-list control group will begin the intervention for the next 8 weeks and activity undergone by participants first randomized into the intervention group will remain under observation.

SUMMARY:
To examine the efficacy of an 8-week exercise training program on functional, cognitive, and emotional health outcomes compared to a no treatment control condition in adults with PASC.

DETAILED DESCRIPTION:
Conduct a randomized control trial with a wait-list control to examine the efficacy of an 8-week exercise training program on functional, cognitive, and emotional health outcomes compared to a no treatment control condition in adults with PASC.

Examine participant compliance (in-person attendance, online engagement) with the 8-week exercise training program including in-person exercise sessions, cognitive performance training, and virtual exercise sessions delivered via a mobile application.

To determine if compliance with the 8-week exercise training program is associated with improvement in functional, cognitive, and emotional health outcomes.

Determine if there is a maintenance effect for individuals randomized into the 8-week exercise training program by comparing their outcomes at the end of the 8-week training exercise program to their outcomes at the end of their trial participation (16 weeks).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Self-reported history of COVID-19 diagnosis
* Self-reported ongoing symptoms of PASC >4 weeks after initial infection

Exclusion Criteria:

* Neuromotor, musculoskeletal, or rheumatoid disorders that are exacerbated by exercise or conditions preventing cooperation
* COVID-19 infection occurring > 6 months prior to screening date
* Contraindications to Symptom-limited Maximal Exercise Testing
* Individuals without access to a device with iOS (apple devices such as iPhone, iPad, MacBook, etc.)
* Patient-reported diagnosis of severe arterial hypertension
* Patient reported metabolic disease
* Patient reported uncontrolled asthma
* Inmates
* Pregnancy
* Patient reported supplemental O2 use
* Presence of beards
* Patient reported diagnosis of claustrophobia
* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Peak Oxygen Consumption (VO2max), mL/min | At first assessment, during week 1.
  Peak oxygen consumption (VO2max) is an indicator of health and fitness. Participants will perform a cardiopulmonary exercise test (CPET) while a metabolic cart measures and calculates their VO2max.
Peak Oxygen Consumption (VO2max), mL/min | At second assessment, during week 11.
  Peak oxygen consumption (VO2max) is an indicator of health and fitness. Participants will perform a cardiopulmonary exercise test (CPET) while a metabolic cart measures and calculates their VO2max.
Peak Oxygen Consumption (VO2max), mL/min | At third assessment, during week 20.
  Peak oxygen consumption (VO2max) is an indicator of health and fitness. Participants will perform a cardiopulmonary exercise test (CPET) while a metabolic cart measures and calculates their VO2max.
Score on Cognitive Function Self-Assessment Scale (CFSS) | At first assessment, during week 1.
  The Cognitive Function Self-Assessment Scale (CFSS) is an 18-item questionnaire designed to self-assess cognitive function. Each question uses a 5-point Likert scale ranging from "never" (0) to "always" (5). The total score is calculated from the mean of the numbers with a lower values indicating a better self-perception of cognitive function and higher values indicating a worse self-perception of cognitive function.
Score on Cognitive Function Self-Assessment Scale (CFSS) | At second assessment, during week 11.
  The Cognitive Function Self-Assessment Scale (CFSS) is an 18-item questionnaire designed to self-assess cognitive function. Each question uses a 5-point Likert scale ranging from "never" (0) to "always" (5). The total score is calculated from the mean of the numbers with a lower values indicating a better self-perception of cognitive function and higher values indicating a worse self-perception of cognitive function.
Score on Cognitive Function Self-Assessment Scale (CFSS) | At third assessment, during week 20.
  The Cognitive Function Self-Assessment Scale (CFSS) is an 18-item questionnaire designed to self-assess cognitive function. Each question uses a 5-point Likert scale ranging from "never" (0) to "always" (5). The total score is calculated from the mean of the numbers with a lower values indicating a better self-perception of cognitive function and higher values indicating a worse self-perception of cognitive function.
Score on PHQ-8 | At first assessment, during week 1.
  The Patient Health Questionnaire (PHQ-8) is an 8-item self-report questionnaire assessing the participant for depression. Each question uses a 4-point scale and the score is determined by the sum of the 8 numbers with higher scores indicating a more severe depression.
Score on PHQ-8 | At second assessment, during week 11.
  The Patient Health Questionnaire (PHQ-8) is an 8-item self-report questionnaire assessing the participant for depression. Each question uses a 4-point Likert scale and the score is determined by the sum of the 8 numbers with higher scores indicating a more severe depression.
Score on PHQ-8 | At third assessment, during week 20.
  The Patient Health Questionnaire (PHQ-8) is an 8-item self-report questionnaire assessing the participant for depression. Each question uses a 4-point Likert scale and the score is determined by the sum of the 8 numbers with higher scores indicating a more severe depression.

SECONDARY OUTCOMES:
Duration, mm:ss | At first assessment, during week 1.
  Total time of test (CPET).
Duration, mm:ss | At second assessment, during week 11.
  Total time of test (CPET).
Duration, mm:ss | At third assessment, during week 20.
  Total time of test (CPET).
Peak VO2 (absolute), mL/min | At first assessment, during week 1.
  Using metabolic cart, absolute peak oxygen consumption will be recorded.
Peak VO2 (absolute), mL/min | At second assessment, during week 11.
  Using metabolic cart, absolute peak oxygen consumption will be recorded.
Peak VO2 (absolute), mL/min | At third assessment, during week 20.
  Using metabolic cart, absolute peak oxygen consumption will be recorded.
Peak VO2 (relative), mL/kg/min | At first assessment, during week 1.
  Using metabolic cart, relative peak oxygen consumption will be recorded.
Peak VO2 (relative), mL/kg/min | At second assessment, during week 11.
  Using metabolic cart, relative peak oxygen consumption will be recorded.
Peak VO2 (relative), mL/kg/min | At third assessment, during week 20.
  Using metabolic cart, relative peak oxygen consumption will be recorded.
Metabolic Equivalents | At first assessment, during week 1.
  Using metabolic cart, metabolic equivalents will be recorded.
Metabolic Equivalents | At second assessment, during week 11.
  Using metabolic cart, metabolic equivalents will be recorded.
Metabolic Equivalents | At third assessment, during week 20.
  Using metabolic cart, metabolic equivalents will be recorded.
Respiratory Exchange Ratio | At first assessment, during week 1.
  Using metabolic cart, respiratory exchange ratio will be recorded.
Respiratory Exchange Ratio | At second assessment, during week 11.
  Using metabolic cart, respiratory exchange ratio will be recorded.
Respiratory Exchange Ratio | At third assessment, during week 20.
  Using metabolic cart, respiratory exchange ratio will be recorded.
VE/VCO2 slope | At first assessment, during week 1.
  Using metabolic cart, VE/VCO2 slope will be recorded.
VE/VCO2 slope | At second assessment, during week 11.
  Using metabolic cart, VE/VCO2 slope will be recorded.
VE/VCO2 slope | At third assessment, during week 20.
  Using metabolic cart, VE/VCO2 slope will be recorded.
Minute Ventilation, L/min | At first assessment, during week 1.
  Using metabolic cart, minute ventilation will be recorded.
Minute Ventilation, L/min | At second assessment, during week 11.
  Using metabolic cart, minute ventilation will be recorded.
Minute Ventilation, L/min | At third assessment, during week 20.
  Using metabolic cart, minute ventilation will be recorded.
Breathing Reserve, % | At first assessment, during week 1.
  Using metabolic cart, breathing reserve will be recorded.
Breathing Reserve, % | At second assessment, during week 11.
  Using metabolic cart, breathing reserve will be recorded.
Breathing Reserve, % | At third assessment, during week 20.
  Using metabolic cart, breathing reserve will be recorded.
Tidal Volume, L | At first assessment, during week 1.
  Using metabolic cart, tidal volume will be recorded.
Tidal Volume, L | At second assessment, during week 11.
  Using metabolic cart, tidal volume will be recorded.
Tidal Volume, L | At third assessment, during week 20.
  Using metabolic cart, tidal volume will be recorded.
Respiratory Frequency, /min | At first assessment, during week 1.
  Using metabolic cart, respiratory frequency will be recorded.
Respiratory Frequency, /min | At second assessment, during week 11.
  Using metabolic cart, respiratory frequency will be recorded.
Respiratory Frequency, /min | At third assessment, during week 20.
  Using metabolic cart, respiratory frequency will be recorded.
Heart Rate, bpm | At first assessment, during week 1.
  Using metabolic cart, heart rate will be recorded.
Heart Rate, bpm | At second assessment, during week 11.
  Using metabolic cart, heart rate will be recorded.
Heart Rate, bpm | At third assessment, during week 20.
  Using metabolic cart, heart rate will be recorded.
Heart Rate Reserve, bpm | At first assessment, during week 1.
  Using metabolic cart, heart rate reserve will be recorded.
Heart Rate Reserve, bpm | At second assessment, during week 11.
  Using metabolic cart, heart rate reserve will be recorded.
Heart Rate Reserve, bpm | At third assessment, during week 20.
  Using metabolic cart, heart rate reserve will be recorded.
Heart Rate Recovery at 1 min, bpm | At first assessment, during week 1.
  Using metabolic cart, heart rate recovery at 1 minute will be recorded.
Heart Rate Recovery at 1 min, bpm | At second assessment, during week 11.
  Using metabolic cart, heart rate recovery at 1 minute will be recorded.
Heart Rate Recovery at 1 min, bpm | At third assessment, during week 20.
  Using metabolic cart, heart rate recovery at 1 minute will be recorded.
VO2/Heart Rate, mL/beat | At first assessment, during week 1.
  Using metabolic cart, VO2/heart rate will be recorded.
VO2/Heart Rate, mL/beat | At second assessment, during week 11.
  Using metabolic cart, VO2/heart rate will be recorded.
VO2/Heart Rate, mL/beat | At third assessment, during week 20.
  Using metabolic cart, VO2/heart rate will be recorded.
VO2 at anaerobic threshold, mL/min | At first assessment, during week 1.
  Using metabolic cart, VO2 at anaerobic threshold will be recorded.
VO2 at anaerobic threshold, mL/min | At second assessment, during week 11.
  Using metabolic cart, VO2 at anaerobic threshold will be recorded.
VO2 at anaerobic threshold, mL/min | At third assessment, during week 20.
  Using metabolic cart, VO2 at anaerobic threshold will be recorded.
PetCO2, mmHg | At first assessment, during week 1.
  Using metabolic cart, end-tidal carbon dioxide pressure (PetCO2) will be recorded.
PetCO2, mmHg | At second assessment, during week 11.
  Using metabolic cart, end-tidal carbon dioxide pressure (PetCO2) will be recorded.
PetCO2, mmHg | At third assessment, during week 20.
  Using metabolic cart, end-tidal carbon dioxide pressure (PetCO2) will be recorded.
PetO2, mmHg | At first assessment, during week 1.
  Using metabolic cart, end-tidal oxygen pressure (PetO2) will be recorded.
PetO2, mmHg | At second assessment, during week 11.
  Using metabolic cart, end-tidal oxygen pressure (PetO2) will be recorded.
PetO2, mmHg | At third assessment, during week 20.
  Using metabolic cart, end-tidal oxygen pressure (PetO2) will be recorded.
VE/VCO2 | At first assessment, during week 1.
  Using metabolic cart, minute ventilation/carbon dioxide production (VE/VCO2) will be recorded.
VE/VCO2 | At second assessment, during week 11.
  Using metabolic cart, minute ventilation/carbon dioxide production (VE/VCO2) will be recorded.
VE/VCO2 | At third assessment, during week 20.
  Using metabolic cart, minute ventilation/carbon dioxide production (VE/VCO2) will be recorded.
Self-Rated Perceived Exertion | At first assessment, during week 1.
  The Borg Rating of Perceived Exertion (6-20) scale will be used during the test to assess subjective exertion. Measured during each stage of the exercise protocol during the cardiopulmonary exercise test. Higher ratings indicating a higher level of exertion.
Self-Rated Perceived Exertion | At second assessment, during week 11.
  The Borg Rating of Perceived Exertion (6-20) scale will be used during the test to assess subjective exertion. Measured during each stage of the exercise protocol during the cardiopulmonary exercise test. Higher ratings indicating a higher level of exertion.
Self-Rated Perceived Exertion | At third assessment, during week 20.
  The Borg Rating of Perceived Exertion (6-20) scale will be used during the test to assess subjective exertion. Measured during each stage of the exercise protocol during the cardiopulmonary exercise test. Higher ratings indicating a higher level of exertion.
Self-Rated Dyspnea | At first assessment, during week 1.
  The Modified Borg Dyspnea Scale (0-10) will be used to assess subjective shortness of breath. Measured during each stage of the exercise protocol during the cardiopulmonary exercise test. Higher values indicating a higher degree of shortness of breath.
Self-Rated Dyspnea | At second assessment, during week 11.
  The Modified Borg Dyspnea Scale (0-10) will be used to assess subjective shortness of breath. Measured during each stage of the exercise protocol during the cardiopulmonary exercise test. Higher values indicating a higher degree of shortness of breath.
Self-Rated Dyspnea | At third assessment, during week 20.
  The Modified Borg Dyspnea Scale (0-10) will be used to assess subjective shortness of breath. Measured during each stage of the exercise protocol during the cardiopulmonary exercise test. Higher values indicating a higher degree of shortness of breath.
Pulse oximetry | At first assessment, during week 1.
  Measured by a pulse oximeter during each stage of the exercise protocol of the cardiopulmonary exercise test on a cycle ergometer.
Pulse oximetry | At second assessment, during week 11.
  Measured by a pulse oximeter during each stage of the exercise protocol of the cardiopulmonary exercise test on a cycle ergometer.
Pulse oximetry | At third assessment, during week 20.
  Measured by a pulse oximeter during each stage of the exercise protocol of the cardiopulmonary exercise test on a cycle ergometer.
Rhythm on electrocardiogram | At first assessment, during week 1.
  Using an electrocardiogram, heart rhythm will be recorded.
Rhythm on electrocardiogram | At second assessment, during week 11.
  Using an electrocardiogram, heart rhythm will be recorded.
Rhythm on electrocardiogram | At third assessment, during week 20.
  Using an electrocardiogram, heart rhythm will be recorded.
Heart Rate Variability (HRV) | Lasting 26 weeks.
  Using the WHOOP 4.0, heart rate variability (HRV) will be calculated and recorded. This will be continuously recorded for 26 weeks.
Respiratory rate | Lasting 26 weeks.
  Using the WHOOP 4.0, respiratory rate will be recorded. This will be continuously recorded for 26 weeks.
Strain | Lasting 26 weeks.
  Using the WHOOP 4.0, strain will be calculated and recorded. This will be continuously recorded for 26 weeks.
Skin temperature, °F | Lasting 26 weeks.
  Using the WHOOP 4.0, skin temperature will be recorded. This will be continuously recorded for 26 weeks.
IPAQ | At first assessment, during week 1.
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) is a 6-item questionnaire assessing how active an individual has been by asking about their activity history. Using the IPAQ, activity history will be recorded.
IPAQ | At second assessment, during week 11.
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) is a 6-item questionnaire assessing how active an individual has been by asking about their activity history. Using the IPAQ, activity history will be recorded.
IPAQ | At third assessment, during week 20.
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) is a 6-item questionnaire assessing how active an individual has been by asking about their activity history. Using the IPAQ, activity history will be recorded.
Motor Speed on CogPT app | At first assessment, during week 1.
  Using the Sports Academy CogPT iPad application, motor speed will be recorded.
Motor Speed on CogPT app | At second assessment, during week 11.
  Using the Sports Academy CogPT iPad application, motor speed will be recorded.
Motor Speed on CogPT app | At third assessment, during week 20.
  Using the Sports Academy CogPT iPad application, motor speed will be recorded.
Reaction Time on CogPT app | At first assessment, during week 1.
  Using the Sports Academy CogPT iPad application, reaction time will be recorded.
Reaction Time on CogPT app | At second assessment, during week 11.
  Using the Sports Academy CogPT iPad application, reaction time will be recorded.
Reaction Time on CogPT app | At third assessment, during week 20.
  Using the Sports Academy CogPT iPad application, reaction time will be recorded.
Reaction Time with No-Go on CogPT app | At first assessment, during week 1.
  Using the Sports Academy CogPT iPad application, reaction time with no-go will be recorded.
Reaction Time with No-Go on CogPT app | At second assessment, during week 11.
  Using the Sports Academy CogPT iPad application, reaction time with no-go will be recorded.
Reaction Time with No-Go on CogPT app | At third assessment, during week 20.
  Using the Sports Academy CogPT iPad application, reaction time with no-go will be recorded.
Dexterity on CogPT app | At first assessment, during week 1.
  Using the Sports Academy CogPT iPad application, dexterity will be recorded.
Dexterity on CogPT app | At second assessment, during week 11.
  Using the Sports Academy CogPT iPad application, dexterity will be recorded.
Dexterity on CogPT app | At third assessment, during week 20.
  Using the Sports Academy CogPT iPad application, dexterity will be recorded.
Inhibition on CogPT app | At first assessment, during week 1.
  Using the Sports Academy CogPT iPad application, inhibition will be recorded.
Inhibition on CogPT app | At second assessment, during week 11.
  Using the Sports Academy CogPT iPad application, inhibition will be recorded.
Inhibition on CogPT app | At third assessment, during week 20.
  Using the Sports Academy CogPT iPad application, inhibition will be recorded.
Dual-Processing on CogPT app | At first assessment, during week 1.
  Using the Sports Academy CogPT iPad application, dual-processing will be recorded.
Dual-Processing on CogPT app | At second assessment, during week 11.
  Using the Sports Academy CogPT application, dual-processing will be recorded.
Dual-Processing on CogPT app | At third assessment, during week 20.
  Using the Sports Academy CogPT iPad application, dual-processing will be recorded.
Working Memory Capacity | At first assessment, during week 1.
  Using the Sports Academy CogPT iPad application, working memory capacity will be recorded.
Working Memory Capacity | At second assessment, during week 11.
  Using the Sports Academy CogPT iPad application, working memory capacity will be recorded.
Working Memory Capacity | At third assessment, during week 20.
  Using the Sports Academy CogPT iPad application, working memory capacity will be recorded.
Sleep duration on WHOOP | Lasting 26 weeks.
  Using the WHOOP 4.0, sleep duration will be recorded. This will be continuously recorded every night for 26 weeks.
Sleep efficiency on WHOOP | Lasting 26 weeks.
  Using the WHOOP 4.0, sleep efficiency will be recorded. This will be continuously recorded every night for 26 weeks.
Sleep stage duration on WHOOP | Lasting 26 weeks.
  Using the WHOOP 4.0, sleep stage duration will be recorded. This will be continuously recorded every night for 26 weeks.
Patient-Reported Outcomes Measurement Information System (PROMIS) | At first assessment, during week 1.
  The Sleep Disturbance-Short Form 4a is derived from the Patient-Reported Outcomes Measurement Information System (PROMIS) and will be used to assess for adult sleep disturbance profiles. It consists of 4-items and is based on a 5-point scale. The sum of each response creates a total raw score. Higher total scores indicate a greater adult sleep disturbance profile. This measure is normed to the US general population.
Patient-Reported Outcomes Measurement Information System (PROMIS) | At second assessment, during week 11.
  The Sleep Disturbance-Short Form 4a is derived from the Patient-Reported Outcomes Measurement Information System (PROMIS) and will be used to assess for adult sleep disturbance profiles. It consists of 4-items and is based on a 5-point scale. The sum of each response creates a total raw score. Higher total scores indicate a greater adult sleep disturbance profile. This measure is normed to the US general population.
Patient-Reported Outcomes Measurement Information System (PROMIS) | At third assessment, during week 20.
  The Sleep Disturbance-Short Form 4a is derived from the Patient-Reported Outcomes Measurement Information System (PROMIS) and will be used to assess for adult sleep disturbance profiles. It consists of 4-items and is based on a 5-point scale. The sum of each response creates a total raw score. Higher total scores indicate a greater adult sleep disturbance profile. This measure is normed to the US general population.
Health Related Quality of Life (EQ-5D) | At first assessment, during week 1.
  Health Related Quality of Life will be assessed using the EuroQol (EQ-5D), a short questionnaire that covers mobility, self-care, activity, pain/discomfort, and anxiety/depression. This tool has shown to be valid, reliable, and responsive in a wide range of conditions and populations.
Health Related Quality of Life (EQ-5D) | At second assessment, during week 11.
  Health Related Quality of Life will be assessed using the EuroQol (EQ-5D), a short questionnaire that covers mobility, self-care, activity, pain/discomfort, and anxiety/depression. This tool has shown to be valid, reliable, and responsive in a wide range of conditions and populations.
Health Related Quality of Life (EQ-5D) | At third assessment, during week 20.
  Health Related Quality of Life will be assessed using the EuroQol (EQ-5D), a short questionnaire that covers mobility, self-care, activity, pain/discomfort, and anxiety/depression. This tool has shown to be valid, reliable, and responsive in a wide range of conditions and populations.
Anxiety (GAD-7) | At first assessment, during week 1.
  Anxiety will be measured using the General Anxiety Disorder-7 (GAD-7). It is a 7-item form, each of which is scored 0 to 3, yielding a 0 to 21 severity score. Higher scores indicating a more severe anxiety. The GAD-7 has shown to be valid, reliable, and sensitive in clinical practice and research.
Anxiety (GAD-7) | At second assessment, during week 11.
  Anxiety will be measured using the General Anxiety Disorder-7 (GAD-7). It is a 7-item form, each of which is scored 0 to 3, yielding a 0 to 21 severity score. Higher scores indicating a more severe anxiety. The GAD-7 has shown to be valid, reliable, and sensitive in clinical practice and research.
Anxiety (GAD-7) | At third assessment, during week 20.
  Anxiety will be measured using the General Anxiety Disorder-7 (GAD-7). It is a 7-item form, each of which is scored 0 to 3, yielding a 0 to 21 severity score. Higher scores indicating a more severe anxiety. The GAD-7 has shown to be valid, reliable, and sensitive in clinical practice and research.
PTSD (LEC-5 and PCL-5) | At first assessment, during week 1.
  Post-traumatic stress disorder (PTSD) symptom severity and trauma history will be assessed using two scales. The Life Events Checklist for DSM-5 (LEC-5) is a 17-item self-report measure designed to screen for traumatic life events. Participants will indicate varying levels of exposure to each type of potentially traumatic event included on a 6-point scale. Additionally, participants will complete the PTSD Check List (PCL-5), a 20-item self-report measure which yields a total symptom severity score of 0-80. Higher scores indicating a greater severity.
PTSD (LEC-5 and PCL-5) | At second assessment, during week 11.
  Post-traumatic stress disorder (PTSD) symptom severity and trauma history will be assessed using two scales. The Life Events Checklist for DSM-5 (LEC-5) is a 17-item self-report measure designed to screen for traumatic life events. Participants will indicate varying levels of exposure to each type of potentially traumatic event included on a 6-point scale. Additionally, participants will complete the PTSD Check List (PCL-5), a 20-item self-report measure which yields a total symptom severity score of 0-80. Higher scores indicating a greater severity.
PTSD (LEC-5 and PCL-5) | At third assessment, during week 20.
  Post-traumatic stress disorder (PTSD) symptom severity and trauma history will be assessed using two scales. The Life Events Checklist for DSM-5 (LEC-5) is a 17-item self-report measure designed to screen for traumatic life events. Participants will indicate varying levels of exposure to each type of potentially traumatic event included on a 6-point scale. Additionally, participants will complete the PTSD Check List (PCL-5), a 20-item self-report measure which yields a total symptom severity score of 0-80. Higher scores indicating a greater severity.
Breathlessness (mMRC) | At first assessment, during week 1.
  Breathlessness will be assessed using the Modified Medical Research Council Dyspnea Scale (mMRC) which is a self-report scale ranging from 0 to 4 commonly used to assess dyspnea during everyday life in patients with pulmonary disease. Higher values indicating a greater condition of dyspnea.
Breathlessness (mMRC) | At second assessment, during week 11.
  Breathlessness will be assessed using the Modified Medical Research Council Dyspnea Scale (mMRC) which is a self-report scale ranging from 0 to 4 commonly used to assess dyspnea during everyday life in patients with pulmonary disease. Higher values indicating a greater condition of dyspnea.
Breathlessness (mMRC) | At third assessment, during week 20.
  Breathlessness will be assessed using the Modified Medical Research Council Dyspnea Scale (mMRC) which is a self-report scale ranging from 0 to 4 commonly used to assess dyspnea during everyday life in patients with pulmonary disease. Higher values indicating a greater condition of dyspnea.
Posttraumatic growth (PTGI) | At first assessment, during week 1.
  Post-traumatic growth will be assessed by the Post-Traumatic Growth Inventory (PTGI), a 21-item scale with possible responses of 0 to 5 assessing positive outcomes after traumatic events. Numerical total score will be obtained and recorded with higher scores indicating a greater degree of change as a result of a crisis.
Posttraumatic growth (PTGI) | At second assessment, during week 11.
  Post-traumatic growth will be assessed by the Post-Traumatic Growth Inventory (PTGI), a 21-item scale with possible responses of 0 to 5 assessing positive outcomes after traumatic events. Numerical total score will be obtained and recorded with higher scores indicating a greater degree of change as a result of a crisis.
Posttraumatic growth (PTGI) | At third assessment, during week 20.
  Post-traumatic growth will be assessed by the Post-Traumatic Growth Inventory (PTGI), a 21-item scale with possible responses of 0 to 5 assessing positive outcomes after traumatic events. Numerical total score will be obtained and recorded with higher scores indicating a greater degree of change as a result of a crisis.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott and White Sports Therapy and Research, Frisco, Texas, United States

IPD SHARING:
Plan to Share IPD: No